CLINICAL TRIAL: NCT01133223
Title: Randomized Clinical Trial Comparing Intravenous Thrombolysis With Thrombectomy by the Penumbra™ System in Patients With Middle Cerebral Artery Stem Occlusion - Pilot Study
Brief Title: Safety and Efficacy of the Penumbra™ System in Acute Middle Cerebral Artery (MCA) Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Lucas Scotta Cabral, Lucas Scotta Cabral, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPPG 09-587
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Stroke
Keywords: Stroke, mecanical thrombectomy
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrombectomy (Active Comparator)
  Interventions: Device: Penumbra™ System
- Usual Care (Active Comparator)
  Interventions: Drug: Recombinant tissue plasminogen activator

INTERVENTIONS:
Device: Penumbra™ System — Patients assigned to the Thrombectomy arm will be conducted to the angio suite. Mechanical thrombectomy will be attempted with the use of the Penumbra™ System, and can be assisted by intraarterial thrombolysis (rTPA up to 20 mg)
  Arms: Thrombectomy
Drug: Recombinant tissue plasminogen activator — Patients assigned to Usual Care arm will be thrombolysed according to the NINDS protocol (rtPA 0,9 mg/kg, 10% IV bolus and remaining in the next hour, up to 90 mg)
  Arms: Usual Care

SUMMARY:
Stroke prognosis is intimately related to reperfusion. Reperfusion in acute setting can be achieved with different strategies - varying from intravenous rtPA from mechanical thrombectomy. Recently, interventional approaches have been gaining attention and playing an increasing role in stroke care. However, no solid scientifical data is available to date. The investigators want do conduct a pilot trial to test if the use of the Penumbra™ System can improve clinical outcomes in a specific stroke setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in acute ischemic stroke protocol
* Up to 3,5h from symptoms onset
* Clinical findings compatible with middle cerebral artery syndrome
* Angiotomographic evidence of proximal middle cerebral artery occlusion

Exclusion Criteria:

* NIHSS < 10
* Overt contraindication to thrombolysis or angiopgraphy
* Disagreement with informed consent term or refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Functional independence (modified Rankin Scale 0-2) | 3 months

SECONDARY OUTCOMES:
Minimal or no disability (modified Rankin Scale 0-1) | 3 months
Overall mortality | 7 days and 3 months
Symptomatic cerebral bleeding rate | 48 hours, 7 days and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Cristina Ouriques Martins, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Background] Ernst R, Pancioli A, Tomsick T, Kissela B, Woo D, Kanter D, Jauch E, Carrozzella J, Spilker J, Broderick J. Combined intravenous and intra-arterial recombinant tissue plasminogen activator in acute ischemic stroke. Stroke. 2000 Nov;31(11):2552-7. doi: 10.1161/01.str.31.11.2552. PMID 11062274
- [Background] Wolpert SM, Bruckmann H, Greenlee R, Wechsler L, Pessin MS, del Zoppo GJ. Neuroradiologic evaluation of patients with acute stroke treated with recombinant tissue plasminogen activator. The rt-PA Acute Stroke Study Group. AJNR Am J Neuroradiol. 1993 Jan-Feb;14(1):3-13. PMID 8427107
- [Background] Mattle HP, Arnold M, Georgiadis D, Baumann C, Nedeltchev K, Benninger D, Remonda L, von Budingen C, Diana A, Pangalu A, Schroth G, Baumgartner RW. Comparison of intraarterial and intravenous thrombolysis for ischemic stroke with hyperdense middle cerebral artery sign. Stroke. 2008 Feb;39(2):379-83. doi: 10.1161/STROKEAHA.107.492348. Epub 2007 Dec 20. PMID 18096842
- [Background] Agarwal P, Kumar S, Hariharan S, Eshkar N, Verro P, Cohen B, Sen S. Hyperdense middle cerebral artery sign: can it be used to select intra-arterial versus intravenous thrombolysis in acute ischemic stroke? Cerebrovasc Dis. 2004;17(2-3):182-90. doi: 10.1159/000075789. Epub 2003 Dec 29. PMID 14707420
- [Background] Noser EA, Shaltoni HM, Hall CE, Alexandrov AV, Garami Z, Cacayorin ED, Song JK, Grotta JC, Campbell MS 3rd. Aggressive mechanical clot disruption: a safe adjunct to thrombolytic therapy in acute stroke? Stroke. 2005 Feb;36(2):292-6. doi: 10.1161/01.STR.0000152331.93770.18. Epub 2004 Dec 29. PMID 15625300
- [Background] Berlis A, Lutsep H, Barnwell S, Norbash A, Wechsler L, Jungreis CA, Woolfenden A, Redekop G, Hartmann M, Schumacher M. Mechanical thrombolysis in acute ischemic stroke with endovascular photoacoustic recanalization. Stroke. 2004 May;35(5):1112-6. doi: 10.1161/01.STR.0000124126.17508.d3. Epub 2004 Mar 11. PMID 15017011
- [Background] Schumacher HC, Meyers PM, Yavagal DR, Harel NY, Elkind MS, Mohr JP, Pile-Spellman J. Endovascular mechanical thrombectomy of an occluded superior division branch of the left MCA for acute cardioembolic stroke. Cardiovasc Intervent Radiol. 2003 May-Jun;26(3):305-8. doi: 10.1007/s00270-003-2719-5. PMID 14562985
- [Background] Kulcsar Z, Bonvin C, Pereira VM, Altrichter S, Yilmaz H, Lovblad KO, Sztajzel R, Rufenacht DA. Penumbra system: a novel mechanical thrombectomy device for large-vessel occlusions in acute stroke. AJNR Am J Neuroradiol. 2010 Apr;31(4):628-33. doi: 10.3174/ajnr.A1924. Epub 2009 Dec 17. PMID 20019113
- [Background] Bose A, Henkes H, Alfke K, Reith W, Mayer TE, Berlis A, Branca V, Sit SP; Penumbra Phase 1 Stroke Trial Investigators. The Penumbra System: a mechanical device for the treatment of acute stroke due to thromboembolism. AJNR Am J Neuroradiol. 2008 Aug;29(7):1409-13. doi: 10.3174/ajnr.A1110. Epub 2008 May 22. PMID 18499798